CLINICAL TRIAL: NCT06102174
Title: AN INTERVENTIONAL, PHASE 1b, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, MULTI-CENTER, DOSE-FINDING STUDY TO EVALUATE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF SISUNATOVIR IN PEDIATRIC PARTICIPANTS UP TO AGE 60 MONTHS WITH RESPIRATORY SYNCYTIAL VIRUS (RSV) LOWER RESPIRATORY TRACT INFECTION (LRTI)
Brief Title: A Study to Learn About the Amount of the Study Medicine (Sisunatovir) in Blood and Its Safety in Infants and Children With Pneumonia Caused by RSV
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study discontinued due to business reasons. There were no safety concerns in the decision to stop study and no changes to sponsor's assessment of the risk-benefit profile for participants who received sisunatovir in the study
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: C5241009; 2023-504425-39-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-06; First posted 2023-10-26 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Lower Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Exercise; sisunatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral or Nasogastric tube (NG)
  Interventions: Drug: Placebo
- Sisunatovir (Active Comparator): Oral or NG tube
  Interventions: Drug: Active

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Active — Sisunatovir
  Other Names: PF-07923568, RV521
  Arms: Sisunatovir

SUMMARY:
The purpose of the study is to learn about the safety and amount of sisunatovir in the blood of infants and children up to age 60 months. These children have Lower Respiratory Tract Infection (LRTI) caused by Respiratory Syncytial Virus (RSV). LRTI is the infection to the lower airways such as lungs.

This study will help inform the amount of sisunatovir to be used in future studies of sisunatovir in children.

This study is seeking for participants who:

* Are 1 day to less than or equal to 60 months of age
* weigh more than or equal to 2.5 kilograms to less than or equal to 23 kilograms.
* Have been tested to have RSV by medical tests.
* show signs of LRTI.

All participants in the study will receive many amounts of sisunatovir or placebo. Placebo is a pill that does not have any medicine in it.

Up to 7 visits are required for the study. Some of these visits include checking participants health over the phone and/or a visit at home.

The study will compare the experiences of infants and children receiving sisunatovir to identify the amount of sisunatovir to be used in future studies in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* 1 day to ≤60 months of age and weight ≥2.5 kg to ≤23 kg
* Positive RSV diagnostic test, antigen or molecular test
* Evidence of Lower Respiratory Tract Infection (LRTI)

Exclusion Criteria:

* Premature infants (gestational age less than 35 weeks) AND <1 year of post-natal age
* Neonates with intrauterine growth restriction
* Expected to receive an antiviral for another viral infection within 10 days of screening
* Suspected or confirmed clinically significant moderate or severe bacterial infection that may interfere with the evaluation of response to the study intervention
* Known to have significant comorbidities that would limit the ability to administer the study intervention or evaluate the safety or clinical response to the study intervention

Ages: 1 Day to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (3):
  - Kaiser Permanente Los Angeles Medical center, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Washington University School of Medicine, St Louis, Missouri
- Japan (4):
  - Kojunkai Daido Hospital, Nagoya, Aichi-ken
  - Nintenkai Kagoshima Children's Hospital, Hioki, Kagoshima-ken
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Osaka City General Hospital, Osaka
- South Africa (2):
  - Monti Clinical Research Centre, Mdantsane, Eastern Cape
  - University of Witwatersrand (WITS) - Vaccines and Infectious Diseases Analytics (VIDA), Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As per plan study was to have 3 cohorts: 1, 2, and 3. Cohorts 1 and 2 was to have further 4 sub-cohorts: A, B, C and D; and Cohort 3 to have sub-cohorts: B, D, E and F. However, due to early termination of study participants were enrolled only in Cohorts 1A, 1B and 1C. No participants were enrolled in Cohort 1D, Cohort 2, and in Cohort 3; hence no results are reported for them. All results are only pertaining to Cohorts 1A, 1B and 1C in this record.
Pre-assignment Details: In this study, participants aged from 1 day to <=60 months received study intervention. Participants of Cohort 1A received study intervention at a low dose level and participants of Cohorts 1B and 1C received study treatment at high dose levels. Cohort 1A had participants of age category 1 (the lowest age category), cohort 1B had participants of age category 2 (medium age category) and cohort 1C had participants of age category 3 (the highest age category).
Groups:
- Cohort 1A: Sisunatovir: Participants of age category 1 were randomized and sisunatovir was administered at low dose level orally or via nasogastric tube for 5 days.
- Cohort 1A: Placebo: Participants of age category 1 were randomized and placebo matched to sisunatovir was administered orally or via nasogastric tube for 5 days.
- Cohort 1B: Sisunatovir: Participants of age category 2 were randomized and sisunatovir was administered at high dose level orally or via nasogastric tube for 5 days.
- Cohort 1B: Placebo: Participants of age category 2 were randomized and placebo matched to sisunatovir was administered orally or via nasogastric tube for 5 days.
- Cohort 1C: Sisunatovir: Participants of age category 3 were randomized and sisunatovir was administered at high dose level orally or via nasogastric tube for 5 days.
- Cohort 1C: Placebo: Participants of age category 3 were randomized and placebo matched to sisunatovir was administered orally or via nasogastric tube for 5 days.
Period: Overall Study
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
Started | 1 | 1 | 2 | 1 | 3 | 2
Completed | 1 | 1 | 2 | 1 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 1 | 3 | 2 | 10
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 1 | 2 | 5
  Male | 0 | 1 | 1 | 1 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2 | 1 | 2 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 1 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 0 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that start on or after the first dose of study intervention, but before the end of the study were flagged as TEAEs. All AEs were included for evaluation.
Time Frame: From start of study intervention on Day 1 up to 28 days after last dose of study intervention (maximum up to 33 days)
Population: Safety population consisted of all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 2
Participants | 0 | 1 | 1 | 1 | 3 | 1

2. Primary Outcome: Number of Participants Who Discontinued From Study Due to TEAEs
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that start on or after the first dose of study intervention, but before the end of the study were flagged as TEAEs.
Time Frame: From start of study intervention on Day 1 up to 28 days after last dose of study intervention (maximum up to 33 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Discontinued From Study Due to Serious TEAEs
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that start on or after the first dose of study intervention, but before the end of the study were flagged as TEAEs. A serious AE (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening experience (immediate risk of death); required inpatient hospitalization or prolongation if existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect; other important event or situation as pre-specified in protocol.
Time Frame: From start of study intervention on Day 1 up to 28 days after last dose of study intervention (maximum up to 33 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, mean cell volume, mean cell hemoglobin & concentration); chemistry: urea and creatinine, estimated glomerular filtration rate (eGFR), gamma-glutamyl transferase (GGT), calcium, sodium, potassium, chloride, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, alkaline phosphatase, albumin, total protein, cystatin C; urinalysis: pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, albumin, creatinine (urine), urine albumin to creatinine ratio. Clinically significant laboratory abnormalities findings were based on investigator discretion.
Time Frame: From start of study intervention on Day 1 up to 28 days after last dose of study intervention (maximum up to 33 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs included systolic and diastolic blood pressure, pulse rate/heart rate, temperature, respiratory rate, and oxygen saturation. Clinically significance vital signs findings were based on investigator discretion.
Time Frame: From start of study intervention on Day 1 up to 28 days after last dose of study intervention (maximum up to 33 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Plasma Concentrations Versus Time Summary of Sisunatovir
Time Frame: Day 3: Pre-dose, T1 and T2 hours post-dose; Day 5: Pre-dose; where T1 is the first analysis time point post-dose while T2 is the second analysis time point post-dose
Population: Pharmacokinetic (PK) concentration set: all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 concentration value can be reported. "Number Analyzed": participants evaluable for specified timepoints, if its value is 0 it means data was missing, PK concentration was not collected at respective timepoint and arm. Data was analyzed and reported only for those arms where participants took sisunatovir, not for placebo arms.
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1B: Sisunatovir | Cohort 1C: Sisunatovir
Number analyzed (Participants) | 1 | 2 | 3
Nanogram per milliliter
  Day 3: Pre-dose: number analyzed (Participants) | 1 | 0 | 1
  Day 3: Pre-dose | NA [NA to NA] — Data was not estimable as PK concentration of the participant was below limit of quantification. |  | 14.0 [14.0 to 14.0]
  Day 3: T1 hours post-dose | 1.9 [1.9 to 1.9] | 19.4 [4.2 to 34.6] | 46.4 [36.0 to 64.6]
  Day 3: T2 hours post-dose | 1.2 [1.2 to 1.2] | 56.3 [51.6 to 60.9] | 34.3 [25.3 to 47.1]
  Day 5: Pre-dose: number analyzed (Participants) | 0 | 2 | 3
  Day 5: Pre-dose |  | 6.3 [5.9 to 6.6] | 12.7 [6.2 to 22.9]

ADVERSE EVENTS:
Time Frame: From start of study intervention on Day 1 up to 28 days after last dose of study intervention (maximum up to 33 days)
Arm/Group | Cohort 1A: Sisunatovir | Cohort 1A: Placebo | Cohort 1B: Sisunatovir | Cohort 1B: Placebo | Cohort 1C: Sisunatovir | Cohort 1C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/1 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 1/2 | 1/1 | 3/3 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A: Sisunatovir (N=1) | Cohort 1A: Placebo (N=1) | Cohort 1B: Sisunatovir (N=2) | Cohort 1B: Placebo (N=1) | Cohort 1C: Sisunatovir (N=3) | Cohort 1C: Placebo (N=2)
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
Sponsor decided to maintain company confidentiality, hence dose strengths, dose frequency, and PK sampling time points have not been disclosed in the record.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT06102174/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT06102174/SAP_001.pdf